CLINICAL TRIAL: NCT01687387
Title: Double-Blind Placebo-Controlled Randomized Phase 2 Study of IPH2102 as Maintenance Treatment in Elderly Patients With Acute Myeloid Leukemia (AML) in First Complete Remission
Brief Title: Efficacy Study of Anti-KIR Monoclonal Antibody as Maintenance Treatment in Acute Myeloid Leukemia (EFFIKIR)
Acronym: EFFIKIR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPH2102-201
Record Dates: First submitted 2012-09-11; First posted 2012-09-18 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2018-09

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — lirilumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IPH2102 at 1 mg/kg (Experimental): lirilumab (IPH2102/BMS986015) at 1 mg/kg
  Interventions: Drug: IPH2102 at 1 mg/kg
- IPH2102 at 0.1 mg/kg (Experimental): lirilumab (IPH2102/BMS986015) at 0.1 mg/kg
  Interventions: Drug: IPH2102 at 0.1 mg/kg; Drug: Placebo (normal saline solution)
- Placebo (Normal saline solution) (Placebo Comparator): Normal saline solution
  Interventions: Drug: Placebo (normal saline solution)

INTERVENTIONS:
Drug: IPH2102 at 0.1 mg/kg — every 3 months
  Other Names: lirilumab/BMS986015
  Arms: IPH2102 at 0.1 mg/kg
Drug: IPH2102 at 1 mg/kg — every 4 weeks
  Other Names: lirilumab/BMS986015
  Arms: IPH2102 at 1 mg/kg
Drug: Placebo (normal saline solution) — every 4 weeks
  Other Names: normal saline solution
  Arms: IPH2102 at 0.1 mg/kg; Placebo (Normal saline solution)

SUMMARY:
Double-Blind Placebo-Controlled Randomized Phase 2 Study evaluating the efficacy of lirilumab (IPH2102/BMS-986015) as Maintenance Treatment administered in elderly patients with Acute Myeloid Leukemia (AML) in first complete remission

ELIGIBILITY:
Inclusion Criteria:

1. Primary or secondary Acute Myeloid Leukemia (AML, defined according to WHO 2008 criteria), in first CR/CRi (according to the revised recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia J Clin Oncol. 2003 Dec 15; 21(24):4642-9 see appendix 19.3) following induction chemotherapy and who received 1 or 2 consolidation cycles. Induction chemotherapy should be performed within 6 months before randomization. Consolidation cycle is defined as any chemotherapy administered within 3 months following CR and including aracytine irrespective of the administered dose(s). A minimum of one and maximum of 2 cycles should be administered before enrollment
2. Patients not eligible for an allogeneic hematopoietic cell transplantation
3. Age 60 to 80
4. ECOG Performance status of 0 or 1
5. Clinical laboratory values at screening

   * Calculated creatinine clearance (according to MDRD) > 60 ml/min/1.73 m2
   * Platelet > 75 x 109/l
   * Hemoglobin ≥ 10 g/dl supported or unsupported by transfusions
   * ANC > 1 x 109/l
   * Total Bilirubin levels ≤ 1.5 ULN
   * ALT and AST ≤ 3 ULN
6. Recovery from acute toxicity of previous anti-tumor therapy
7. Male patients who accept and are able to use contraception methods recognized as highly effective.
8. Signed informed consent prior to any protocol specific procedure.

Exclusion Criteria:

1. Acute Promyelocytic Leukemia with t (15; 17), or its molecular equivalents (PML-RARA)
2. Favorable risk AML corresponding defined as t(8;21) or inv (16) and t(16;16) and their molecular equivalents (AML-ETO and CBFB-MYH11)
3. Last consolidation completed more than 3 months prior to first dosing
4. Concomitant treatment by chemotherapy, immunotherapy or by systemic corticosteroids
5. Within 28 days prior to first dosing: chemotherapy or systemic corticosteroid treatment
6. History of allogeneic hematopoietic cell transplantation or solid organ transplantation
7. History of high dose chemotherapy with autologous hematopoietic transplantation performed as treatment for AML
8. Use of any investigational agent within 2 months prior to the first dosing
9. Use of growth factors (G- or GM-CSF or EPO) within 28 days prior to first dosing
10. Any irradiation within the last 3 months except for analgesic intent
11. Intermittent or continuous renal replacement therapy
12. Abnormal cardiac status with any of the following

    * Ejection fraction (measured by ultra-sound or radionuclide imaging) <50%
    * Myocardial infarction within the previous 6 months
    * QTc ≥ 480 ms (Bazett's).
13. Current active infectious disease or positive serology for HIV, and/or HCV with detectable viremia and/ or HBV with positive Hbs Antigen and/or negative anti Hbs Antibody
14. Auto-immune disease:

    * Which currently or previously required systemic immunosuppressive or immuno-modulatory therapy (including corticosteroids administered by systemic route)
    * And/or has substantial probability to cause an irreversible injury to any tissue
    * And/or is recent or unstable or has substantial risk to progress and cause severe complications.
15. Serious concurrent uncontrolled medical disorder
16. History of another malignancy (apart from myelodysplastic syndromes, basal cell carcinoma of the skin, or in situ cervix carcinoma) except if free of disease for ≥ 3 years
17. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2012-10; Primary Completion 2016-11-17 (Actual); Study Completion 2016-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Vey, MD, Principal Investigator — Institut Paoli Calmettes Marseille France; Hervé Dombret, MD, Study Chair — ALFA cooperative Group; Norbert Ifrah, MD, Study Chair — GOELAMS Cooperative Group
Locations (43):
- France (43):
  - CHU d'Amiens, Amiens
  - CHU Angers, Angers
  - Centre hospitalier Victor Dupouy, Argenteuil
  - Centre hospitalier de la côte Basque, Bayonne
  - CHU de Besançon, Besançon
  - CHG de Béziers, Béziers
  - CH de Blois, Blois
  - Hôpital Avicenne, Bobigny
  - Hôpital Morvan CHU Brest, Brest
  - CH René Dubos, Cergy-Pontoise
  - Hôpital Militaire Percy, Clamart
  - CHU Estaing, Clermont-Ferrand
  - Centre hospitalier sud francilien, Corbeil-Essonnes
  - Hôpital Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - Centre Hospitalier de Versailles, Le Chesnay
  - Hôpital Claude Huriez, Lille
  - CHU de Limoges, Limoges
  - Institut Paoli - Calmettes, Marseille
  - CH de Meaux, Meaux
  - CHU Saint Eloi, Montpellier
  - Centre Hospitalier de Mulhouse, Mulhouse
  - CHU de Nantes, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU Caremeau, Nîmes
  - CHR d'Orléans, Orléans
  - Hôpital Saint-Louis, Paris
  - Hôpital Saint-Antoine, Paris
  - Hôpital Necker, Paris
  - CH Saint-Jean, Perpignan
  - CHU de Bordeaux - Hôpital Haut-Lévêque, Pessac
  - Centre hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - CHR d'Annecy, Pringy
  - CHU de Reims, Reims
  - Centre Henri Becquerel, Rouen
  - Centre René Huguenin, Saint-Cloud
  - CH Saint-Quentin, Saint-Quentin
  - Hôpital Haute Pierre et Hôpital Civil, Strasbourg
  - CHU Purpan, Toulouse
  - CH Valenciennes, Valenciennes
  - CHU de Nancy Hôpitaux de Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 169 patients were screened and 152 patients were randomized and treated in France
Period: Overall Study
Arm/Group | IPH2102 at 1 mg/kg | IPH2102 at 0.1 mg/kg | Placebo (Normal Saline Solution)
Started | 51 | 50 | 51
Completed | 10 | 12 | 13
Not Completed | 41 | 38 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IPH2102 at 1 mg/kg | IPH2102 at 0.1 mg/kg | Placebo (Normal Saline Solution) | Total
Number analyzed (Participants) | 51 | 50 | 51 | 152
Age, Continuous [Median (Full Range); unit: years] | 70 [60 to 80] | 70 [60 to 80] | 68 [60 to 77] | 70 [60 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 16 | 17 | 61
  Male | 23 | 34 | 34 | 91
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 51 | 50 | 51 | 152

OUTCOME MEASURES:

1. Primary Outcome: Leukemia-Free Survival
Time Frame: from date of randomization until the date of first documented relapse, assessed up to 48 months
Measure: Median (95% Confidence Interval); unit: MONTHS
Arm/Group | IPH2102 at 1 mg/kg | IPH2102 at 0.1 mg/kg | Placebo (Normal Saline Solution)
Number analyzed (Participants) | 51 | 50 | 51
MONTHS | 6.7 [2.9 to 14.8] | 17.6 [11.2 to 25] | 13.9 [7.9 to 27.9]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of Participants with Adverse Events based on full physical examination each treatment visit and collection of AEs
Time Frame: from the time of patient signing the consent form until 28 days after the last administration, or until the patient's last study visit, up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | IPH2102 at 1 mg/kg | IPH2102 at 0.1 mg/kg | Placebo (Normal Saline Solution)
Number analyzed (Participants) | 51 | 50 | 51
Participants | 43 | 49 | 47

ADVERSE EVENTS:
Time Frame: AEs and SAEs will be collected throughout the study from the time of patient signing the consent form until 28 days after the last administration, or until the patient's last study visit
Arm/Group | IPH2102 at 1 mg/kg | IPH2102 at 0.1 mg/kg | Placebo (Normal Saline Solution)
All-Cause Mortality (participants affected / at risk) | 32/51 | 26/50 | 23/51
Serious Adverse Events (participants affected / at risk) | 12/51 | 17/50 | 11/51
Other Adverse Events (participants affected / at risk) | 38/51 | 48/50 | 43/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IPH2102 at 1 mg/kg (N=51) | IPH2102 at 0.1 mg/kg (N=50) | Placebo (Normal Saline Solution) (N=51)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Chorioretinal disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Injury corneal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Biopsy spleen (Investigations) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 2 (2)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Myxofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory therapy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IPH2102 at 1 mg/kg (N=51) | IPH2102 at 0.1 mg/kg (N=50) | Placebo (Normal Saline Solution) (N=51)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 5 (5) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 4 (9) | 4 (5) | 5 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (9) | 7 (11) | 3 (4)
Conjunctivitis (Eye disorders) | 3 (3) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (4) | 2 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (4) | 5 (5) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 6 (6) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (3) | 6 (6) | 3 (3)
Asthenia (General disorders) | 14 (20) | 14 (19) | 14 (22)
Chest pain (General disorders) | 1 (1) | 4 (4) | 2 (2)
Chills (General disorders) | 4 (5) | 3 (4) | 1 (2)
Fatigue (General disorders) | 5 (5) | 2 (2) | 3 (4)
Influenza like illness (General disorders) | 2 (2) | 4 (5) | 5 (9)
Oedema peripheral (General disorders) | 1 (1) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 6 (6) | 3 (3) | 5 (5)
Bronchitis (Infections and infestations) | 6 (9) | 17 (20) | 14 (15)
Gastroenteritis (Infections and infestations) | 1 (1) | 4 (5) | 3 (4)
Nasopharyngitis (Infections and infestations) | 2 (2) | 6 (6) | 6 (7)
Oral herpes (Infections and infestations) | 0 (0) | 2 (2) | 3 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (4) | 2 (8) | 5 (7)
Lipase increased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Weight increased (Investigations) | 1 (1) | 5 (6) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6) | 5 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (7) | 7 (8)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 5 (6)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 6 (6)
Headache (Nervous system disorders) | 8 (9) | 4 (9) | 3 (5)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 3 (4) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 6 (9) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 3 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (9) | 10 (11) | 7 (12)
Hypertension (Vascular disorders) | 2 (2) | 5 (6) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No